CLINICAL TRIAL: NCT04060992
Title: Can Hormonal Effects of the Oral Gonadotropin Releasing Hormone (GnRH) Antagonist Withstand When Administered at Different Points in the Menstrual Cycle?
Brief Title: Hormonal Effects of the Oral Gonadotropin Releasing Hormone (GnRH) Antagonist at Different Periods of the Menstrual Cycle
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Frank Stanczyk, Research Progessor of Obstetrics & Gynecology, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APP-19-02687
Record Dates: First submitted 2019-08-07; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Ovulation; Failure or Lack of
MeSH Terms: conditions — Anovulation | interventions — elagolix; Tablets

STUDY DESIGN:
Intervention Model Description: Observational study design, prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early Follicular Phase (Experimental): Women enrolled will be anywhere from cycle day 1 through 5 of their menstrual cycle and take elagolix 200mg oral tablet BID for 3 days total.
  Interventions: Drug: Elagolix 200 MG Oral Tablet [Orilissa]
- Late Follicular Phase (Active Comparator): Women enrolled will be anywhere from cycle day 8 through 13 of their menstrual cycle and take elagolix 200mg oral tablet BID for 3 days total.
  Interventions: Drug: Elagolix 200 MG Oral Tablet [Orilissa]
- Luteal Phase (Active Comparator): Women enrolled will be anywhere from cycle day 21 through cycle day 26 of their menstrual cycle and take elagolix 200mg oral tablet BID for 3 days total.
  Interventions: Drug: Elagolix 200 MG Oral Tablet [Orilissa]

INTERVENTIONS:
Drug: Elagolix 200 MG Oral Tablet [Orilissa] — oral tablet given twice daily

SUMMARY:
The purpose of this study is twofold: First, to see if elagolix can suppress gonadotropin and ovarian hormones in the short-term period, when only administered for a 72-hour period. If elagolix effectively suppresses gonadotropin and ovarian hormones in a timely manner, it could be used to alter aspects of the menstrual cycle, depending on when administered. Second, is there a window for when elagolix functions best? While other studies initiate elagolix at the start of a woman's menstrual cycle, investigators of this study want to determine if administering elagolix at various points in a woman's menstrual cycle alters its ability to suppress gonadal and ovarian hormones.

DETAILED DESCRIPTION:
Gonadotropin-releasing hormone (GnRH) and its analogs have been utilized in clinical medicine since the early 1970s. The GnRH analog is more potent with a longer half-life than native GnRH. When administered continuously rather than in a more physiologic pulsatile manner, the initial stimulation of pituitary gonadotrophs is followed by pituitary desensitization1,2. This ultimately leads to inhibition of the pituitary-gonadal axis. This downregulation facilitates the use of GnRH agonists for the treatment of various medical conditions, including precocious puberty, endometriosis, uterine leiomyomata, prostate cancer, and assisted reproductive technology (ART)1,2.

Like GnRH agonists, antagonists of GnRH have proven to efficiently suppress pituitary and ovarian hormone production. However, unlike the agonist, the GnRH-antagonist competitively binds to the GnRH-receptor1,2. The antagonist bypasses the initial flare effect and does not require the initial period of administration for pituitary desensitization of GnRH receptors. As a result, there is rapid prevention of gonadotropin secretion and antagonist effect on the ovary1-4.

In addition to the enhanced efficiency of using a GnRH-antagonist, it has shown to be more tolerable with fewer side effects when compared to the older GnRH agonist1-5. Particularly in ART, GnRH agonists are associated with hot flashes, ovarian cyst formation, and ovarian hyperstimulation syndrome (OHSS)6. Conversely, GnRH antagonists have been shown to significantly reduce the incidence of OHSS, and are not associated with cyst development or hot flashes6. It is important to note that in ART literature, administration of a GnRH-antagonist has been via a subcutaneous injection, formulated as ganirelix, detirelix or cetrotide3-5.

Fluker et al investigated the impact of the subcutaneous GnRH-antagonist on gonadotropin and ovarian hormone production when administered at different points of the menstrual cycle: mid-follicular phase, preovulatory phase, and early luteal phase5. Investigators found that the GnRH-antagonist successfully suppressed gonadotropin hormones irrespective of phase of menstrual cycle. Suppression of ovarian hormones, and particularly suppression of the LH surge, was evident only when the GnRH-antagonist administered in mid-follicular and early luteal phases5.

In an effort to avoid a subcutaneous injection and ease patient administration, an oral GnRH-antagonist has recently been developed: Elagolix. Research has shown that elagolix similarly suppresses gonadotropin and ovarian hormones compared to its injectable formulary7.

Ng et al investigated the pharmacokinetics of elagolix over a 21-day period, while also investigating elagolix's suppression of gonadotropic and ovarian hormones at varying doses when administered during a natural menstrual cycle7. Time to maximum concentration of elagolix was 1.0-1.5 hours, with a half-life of about 4-6 hours. While maximum suppression of follicle stimulating hormone (FSH) and LH occurred in all doses administered, maximum suppression was seen in the elagolix 300mg BID and 400mg BID groups. Rebound to baseline FSH and LH was evident within 24-48 hours from last dose of elagolix. Maximum estradiol suppression was seen when administered at 200mg BID or higher doses, and maximum progesterone suppression was seen in all doses 100mg BID or higher. While elagolix was administered for a 21-day period, the greatest decrease in gonadotropin and ovarian hormone levels was seen in the first three days of administration at any dose7.

Thus far, the Federal Drug Administration (FDA) has approved elagolix for the management of moderate to severe pain associated with endometriosis. Approved regimens include one 150mg tablet once daily or one 200mg tablet twice daily7-10. Like the injectable GnRH antagonist, the oral GnRH antagonist efficiently manages pain symptoms in endometriosis via suppression of estrogen secretion. Estrogen is thought to play a role in the pathophysiology of endometriosis via its stimulatory effects on the endometrium and its stimulatory effects on a woman's inflammatory milieu, both at the local and systemic level10.

While elagolix has been proven to effectively suppress gonadotropin and ovarian hormones, like the injectable GnRH antagonists, elagolix has yet to be used in conditions other than endometriosis, such as in cases of ART7. More specifically, the impact of elagolix in the short-term period for cases of COH has yet to be studied.

Subjectively looking at Ng et al's data, there are sharp declines in FSH, LH, estradiol, and progesterone within the first three days of administering elagolix, and these concentrations continue to decline, but at a less steep slope, from days 4 through day 21 of administration7. It appears that the first three days are crucial to hormonal suppression7.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers from USC Fertility
* Documented ovulation with a serum mid-luteal progesterone ≥3pg/mL
* Ovulatory with a 24-35-day cycle
* Ages 18-39
* Body Mass Index (BMI) 18.1-30.0kg/m2
* Consistent condom use for contraception
* Not desiring or seeking pregnancy

Exclusion Criteria:

* Allergy to injectable or oral GnRH-antagonist
* FSH ≥ 10 IU/L or LH ≥ 10 IU/L in early follicular phase iii. Known liver disease iv. Known osteoporosis v. Pregnancy vi. Current use of drugs metabolized by the liver enzyme CYP3A, specifically ketoconazole, rifampin, digoxin, oral midazolam, or rosuvastatin.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Suppression of gonadotropin and pituitary hormones as measured by hormonal assay status post short-term administration of elagolix | measured over 4 days
  Measure serum concentrations of follicle stimulation hormone (FSH), luteinizing hormone (LH), estradiol, progesterone at baseline and throughout three-day course of elagolix

SECONDARY OUTCOMES:
Time interval to next menses | up to 4 weeks
  Calculate number of days from elagolix consumption to next menses

IPD SHARING:
Plan to Share IPD: No
No, data will not be available to other researchers. At the study completion, all patient data will be destroyed in the HIPAA compliant manner.

REFERENCES:
- [Result] Kumar P, Sharma A. Gonadotropin-releasing hormone analogs: Understanding advantages and limitations. J Hum Reprod Sci. 2014 Jul;7(3):170-4. doi: 10.4103/0974-1208.142476. PMID 25395741
- [Result] Andreyko JL, Marshall LA, Dumesic DA, Jaffe RB. Therapeutic uses of gonadotropin-releasing hormone analogs. Obstet Gynecol Surv. 1987 Jan;42(1):1-21. PMID 3543765
- [Result] Fluker M, Grifo J, Leader A, Levy M, Meldrum D, Muasher SJ, Rinehart J, Rosenwaks Z, Scott RT Jr, Schoolcraft W, Shapiro DB; North American Ganirelix Study Group. Efficacy and safety of ganirelix acetate versus leuprolide acetate in women undergoing controlled ovarian hyperstimulation. Fertil Steril. 2001 Jan;75(1):38-45. doi: 10.1016/s0015-0282(00)01638-1. PMID 11163814
- [Result] Garcia-Velasco JA, Isaza V, Vidal C, Landazabal A, Remohi J, Simon C, Pellicer A. Human ovarian steroid secretion in vivo: effects of GnRH agonist versus antagonist (cetrorelix). Hum Reprod. 2001 Dec;16(12):2533-9. doi: 10.1093/humrep/16.12.2533. PMID 11726570
- [Result] Fluker MR, Marshall LA, Monroe SE, Jaffe RB. Variable ovarian response to gonadotropin-releasing hormone antagonist-induced gonadotropin deprivation during different phases of the menstrual cycle. J Clin Endocrinol Metab. 1991 Apr;72(4):912-9. doi: 10.1210/jcem-72-4-912. PMID 2005218
- [Result] Depalo R, Jayakrishan K, Garruti G, Totaro I, Panzarino M, Giorgino F, Selvaggi LE. GnRH agonist versus GnRH antagonist in in vitro fertilization and embryo transfer (IVF/ET). Reprod Biol Endocrinol. 2012 Apr 13;10:26. doi: 10.1186/1477-7827-10-26. PMID 22500852
- [Result] Ng J, Chwalisz K, Carter DC, Klein CE. Dose-Dependent Suppression of Gonadotropins and Ovarian Hormones by Elagolix in Healthy Premenopausal Women. J Clin Endocrinol Metab. 2017 May 1;102(5):1683-1691. doi: 10.1210/jc.2016-3845. PMID 28323948
- [Result] Elagolix (Orilissa)--an oral GnRH antagonist for endometriosis pain. Med Lett Drugs Ther. 2018 Sep 24;60(1556):158-160. No abstract available. PMID 30383729
- [Result] Surrey E, Taylor HS, Giudice L, Lessey BA, Abrao MS, Archer DF, Diamond MP, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Singh SS, Rechberger T, Agarwal SK, Duan WR, Schwefel B, Thomas JW, Peloso PM, Ng J, Soliman AM, Chwalisz K. Long-Term Outcomes of Elagolix in Women With Endometriosis: Results From Two Extension Studies. Obstet Gynecol. 2018 Jul;132(1):147-160. doi: 10.1097/AOG.0000000000002675. PMID 29889764
- [Result] Taylor HS, Giudice LC, Lessey BA, Abrao MS, Kotarski J, Archer DF, Diamond MP, Surrey E, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Rowan JP, Duan WR, Ng J, Schwefel B, Thomas JW, Jain RI, Chwalisz K. Treatment of Endometriosis-Associated Pain with Elagolix, an Oral GnRH Antagonist. N Engl J Med. 2017 Jul 6;377(1):28-40. doi: 10.1056/NEJMoa1700089. Epub 2017 May 19. PMID 28525302
- [Derived] Danis RB, Sriprasert I, Stanczyk FZ, Paulson RJ, Winer SA, Ho JR. Does timing matter when initiating elagolix in a natural menstrual cycle? F S Rep. 2021 May 31;2(3):308-313. doi: 10.1016/j.xfre.2021.05.009. eCollection 2021 Sep. PMID 34553156